CLINICAL TRIAL: NCT07368556
Title: The Effect of a Nursing Care Program Based on Human Caring Theory on Self-Esteem, Coping, and Self-Compassion in Adolescents With Self-Harm
Brief Title: The Impact of a Nursing Care Program Based on Human Caring Theory on Adolescents With Self-harm
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Hilal Kara, Registered Nurse, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AU-SBE-HK-01
Record Dates: First submitted 2026-01-20; First posted 2026-01-26 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Self Harm
Keywords: self harm; adolescent; psychiatric nursing; randomized controlled trial
MeSH Terms: conditions — Self-Injurious Behavior

STUDY DESIGN:
Intervention Model Description: It is a randomized controlled, single-blind experimental study. There is an experimental and control group
Who Masked: Participant
Masking Description: For the randomization process, the distribution obtained from the Statistical Analysis System (SAS) statistical program will be placed in sealed envelopes by someone other than the researcher, and the envelopes will be numbered. Adolescents who meet the inclusion criteria and agree to participate in the study will be assigned to either the intervention group or the control group after the envelopes are opened. This ensures a one-way blinding process, preventing adolescents diagnosed with self-harm from knowing whether they are in the intervention or control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group receiving Nursing Care Program based on Human Caring Theory (Experimental): In addition to routine treatment and follow-up at the Child and Adolescent Mental Health and Diseases Outpatient Clinic, the Human Caring Theory-Based Nursing Care Program will be implemented face-to-face and individually through therapeutic interviews.
  Interventions: Behavioral: Group receiving Nursing Care Program based on Human Caring Theory
- Group receiving routine treatment and follow-up at the polyclinic. (Active Comparator): The control group will receive only routine treatment and follow-up at the Child and Adolescent Mental Health and Diseases Outpatient Clinic.
  Interventions: Behavioral: Group receiving routine treatment and follow-up at the polyclinic.

INTERVENTIONS:
Behavioral: Group receiving Nursing Care Program based on Human Caring Theory — Adolescents who can be included in the study are determined by interviewing the group of physicians working at the Child and Adolescent Mental Health and Diseases Outpatient Clinic of Antalya City Hospital. Providing verbal information about the research to adolescents and parents/guardians, obtaining written consent from adolescents and parents/guardians who agree to participate in the research, administering the measurement tools,implementing the Human Caring Theory-Based Nursing Care Program for a total of six weeks, once a week, re-administering the measurement tools, conducting a follow-up measurement after six weeks,terminating the interview.
  Arms: Group receiving Nursing Care Program based on Human Caring Theory
Behavioral: Group receiving routine treatment and follow-up at the polyclinic. — Adolescents who can be included in the study are determined by interviewing the group of physicians working at the Child and Adolescent Mental Health and Diseases Outpatient Clinic of Antalya City Hospital. Providing verbal information about the research to adolescents and parents/guardians, obtaining written consent from adolescents and parents/guardians who agree to participate in the research, administering the measurement tools, application of measurement tools after six weeks, follow-up measurement after six weeks, terminating the interview.
  Arms: Group receiving routine treatment and follow-up at the polyclinic.

SUMMARY:
The aim of this study is to examine the effect of a Nursing Care Program based on Human Caring Theory on self-esteem, coping, and self-compassion in adolescents exhibiting self-harming behavior.

Hypotheses of the research:

H1-a: The self-esteem level of adolescents exhibiting self-harm in the intervention group that received the Human Caring Theory-Based Nursing Care Program differed significantly from the control group.

H1-b: The self-compassion level of adolescents exhibiting self-harm in the intervention group that received the Human Caring Theory-Based Nursing Care Program differed significantly from the control group.

H1-c: The coping level of adolescents exhibiting self-harm in the intervention group that received the Human Caring Theory-Based Nursing Care Program differed significantly from the control group.

This study is a randomized, controlled, single-blind experimental design. It will be conducted between January 2026 and March 2027 at the Child and Adolescent Mental Health and Diseases Outpatient Clinic of Antalya City Hospital with 54 adolescents (27 in the intervention group and 27 in the control group) who meet the inclusion criteria. The Human Caring Theory-Based Nursing Care Program will be applied individually and face-to-face to adolescents in the intervention group through structured therapeutic interviews. Data will be collected using a Personal Information Form, the Inventory of Statements About Self-injury, the Rosenberg Self-Esteem Scale, the Coping Scale for Adolescents, and the Short Form of the Self-Compassion Scale. Data analysis will be performed using the Statistical Package for Social Science (SPSS) 31.0 software package. It is believed that the Human Caring Theory-Based Nursing Care Program may be effective in improving self-esteem, self-compassion, and coping skills in adolescents exhibiting self-harm behavior.

DETAILED DESCRIPTION:
Self-harm is when an individual injures or harms themselves in order to cope with or express emotional distress and confusion. Examples of self-harm include attempting to poison oneself by overdosing on drugs or harmful substances, cutting and scratching the skin, self-burning, and punching oneself. Systematic reviews and meta-analyses of various countries, including Turkey, have found that self-harm behavior ranges from 16% to 17.7% and is particularly high among adolescents. Furthermore, systematic reviews and meta-analyses indicate that self-harm is more common in adolescent girls than in adolescent boys, and is higher in Asia. Umbrella reviews, systematic reviews, and meta-analyses show that many factors influence suicidal and self-harm. Self-esteem, self-compassion, and coping skills are some of the risk factors for self-harm.

Self-harm is a strong predictor of suicide attempts, is repetitive, and is one of the leading causes of death. Early intervention for self-harm can reduce the risk of suicide and death later in life. It is emphasized that planned interventions for self-harm should include alternative behavioral skills and problem-solving strategies, address the individual's strengths in collaboration, utilize individualized coping methods and self-care approaches, and be individualized, structured, and limited in duration. Human Caring Theory adopts the approach that each individual is unique and requires a holistic approach, that treatment is possible only with the individual's participation, and that the individual cannot be considered separately from their environment. Accordingly, it may be appropriate and effective for psychiatric nurses caring for adolescents exhibiting self-harm to base their care processes on Human Caring Theory. A review of the literature reveals that studies in nursing with adolescents based on Human Caring Theory are limited, and additionally, no experimental studies with individuals exhibiting self-harm behavior have been found. It is thought that a nursing care program based on the Human Caring Theory can contribute to the development of coping skills, self-compassion, and self-esteem in adolescents exhibiting self-harm, and can also reduce this behavior. The study suggests that this approach may be effective in protecting adolescents with self-harm from the risk of suicidal behavior and life-threatening risks associated with self-harm, and in maintaining their healthy development.

ELIGIBILITY:
Inclusion Criteria:

The study will include adolescents who:

* are aged 14-18 years,
* volunteer to participate in the study, and
* have self-harm according to Diagnostic and Statistical Manual of Mental Disorders (DSM-5) diagnostic criteria.

Exclusion Criteria:

* Adolescents with speech, hearing, comprehension, or visual impairments, as well as those receiving psychosocial support during the research process, will not be included in the study.

Sampling Exclusion Criteria:

* Adolescents who did not participate in all interviews
* Were admitted to the Child and Adolescent Psychiatry clinic for treatment during the research process,
* Did not wish to continue participating in the interviews will be excluded from the study.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 54 (Estimated)
Dates: Start 2026-01-29 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Rosenberg Self Esteem Scale (RSE) | six weeks
  1st, 2nd, and 3rd questions; 4th and 5th questions; and 9th and 10th questions are evaluated together.
  If a respondent receives points on any two of the first three questions (2 out of 3), they receive one point from this set.
  If they select one of the options that receives a point in either the 4th or 5th question, they also receive one point from this set.
  The 9th and 10th questions are evaluated in the same way as the 4th and 5th questions.
  The 6th, 7th, and 8th questions are each scored individually. Thus, when a respondent receives points from all question sets, the maximum possible total score is 6.
The Short Form of Self-Compassion Questionnaire | six weeks
  The Short Form of the Self-Compassion Scale can be administered to middle school and high school students.
  Items 1, 4, 8, 9, 10, and 11 on the scale are reverse-coded. As the total score obtained from the scale increases, the level of self-compassion also increases.
  During the adaptation of the scale into Turkish, one item was removed.
Coping Scale for Adolescents (CSA) | six weeks
  The scale consists of 11 items. Items 3, 6, 8, and 10 are related to active coping. Items 1, 2, 9, and 11 are related to avoidance coping. Items 4, 5, and 7 are related to negative coping.
  Each subscale score is obtained by summing the scores of the relevant items. The possible score range is 0-12 for active coping and avoidance coping, and 0-9 for negative coping. Higher scores on the scale indicate more frequent use of the corresponding coping approach.

CONTACTS AND LOCATIONS:
Overall Officials: Dudu KARAKAYA, PhD, Study Director — Akdeniz University; Hilal KARA, MSN, Principal Investigator — Akdeniz University
Locations (1):
- Antalya City Hospital, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No